CLINICAL TRIAL: NCT04729439
Title: Development of a Technology-Enhanced Executive Functioning Skills Intervention for Adolescents With ADHD
Brief Title: Technology-Enhanced Executive Functioning Intervention for ADHD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Melissa Dvorsky, Psychologist, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO#00014877
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder; Attention Deficit Disorder; ADD; ADHD Predominantly Inattentive Type; ADHD - Combined Type; ADHD, Predominantly Hyperactive - Impulsive; Attention-Deficit Disorder in Adolescence; Attention-Deficit Hyperactivity Disorder Symptoms; Attention-Deficit Hyperactivity Disorder
Keywords: ADHD; Attention-Deficit/Hyperactivity Disorder; Executive Functioning
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — ALPL protein, human; Methods

STUDY DESIGN:
Intervention Model Description: A preliminary feasibility effectiveness trial comparing two groups: (1) organizational/behavioral skills intervention augmented with digital health application and (2) organizational/behavioral skills intervention only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Organizational/behavioral intervention + digital health tool (Experimental): Participants will receive sixteen 30-minute sessions of the organizational/behavioral skills intervention (i.e., Homework Organization and Planning Skills [HOPS]) plus the online digital health application during treatment
  Interventions: Behavioral: Homework Organization and Planning Skills (HOPS) Intervention; Device: Digital Health Application (Online Platform) for Encouraging Skills Practice
- Organizational/behavioral intervention only (Active Comparator): Participants will receive sixteen 30-minute sessions of the organizational/behavioral skills intervention (i.e., Homework Organization and Planning Skills [HOPS]) only, without the online digital health application during treatment
  Interventions: Behavioral: Homework Organization and Planning Skills (HOPS) Intervention

INTERVENTIONS:
Behavioral: Homework Organization and Planning Skills (HOPS) Intervention — A behavioral/organizational skills intervention focused on improving adolescents' homework, organization, and planning skills
Device: Digital Health Application (Online Platform) for Encouraging Skills Practice — This online platform can be used on participants' personal devices including laptops, phones, tablets, or other computers and is designed to encourage adolescent's skills practice, monitor and reward treatment progress, and optimize motivation in treatment
  Other Names: Advanced Tools for Organization Management
  Arms: Organizational/behavioral intervention + digital health tool

SUMMARY:
This study develops and refines an online platform that will support clinician-directed behavioral and organizational skills intervention for adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD) with input guided from key stakeholders during focus groups and interviews (phase 1), extended usability testing (phase 2), and a pilot randomized trial (phase 3) of the online tool used in conjunction with an organizational skills intervention.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is one of the most common childhood mental health disorders, affecting 7-9% of youth and leading to substantial impairment in adolescence. Despite evidence suggesting that behavioral interventions are efficacious, 41-60% of adolescents receiving behavioral treatment show little to no improvement and skills are rarely generalized beyond treatment sessions. Lack of adolescent motivation and engagement, between-session skills use, reward saliency, and family involvement are key contributors to these limited effects. Mobile digital health strategies and gamification techniques offer transformative opportunities for overcoming the barriers of evidence-based treatments specific to ADHD by using interactive tools to reinforce in-vivo skill practice, providing opportunities for immediate reinforcement, and motivating adolescents with digital rewards. The goal of this proposal is to develop and evaluate an online platform tool that will support clinician-directed behavioral treatment for adolescents with ADHD by improving executive functioning skills acquisition and utilization, providing in-vivo skills reinforcement, and monitoring adolescents' skill utilization. This study will use an empirically supported intervention specifically designed to address the domains of impairment frequently experienced by adolescents with ADHD. This study will use an iterative stakeholder-centered design to develop, refine, and preliminarily test a scalable digital health tool, applied as an adjunct to behavioral treatment for adolescents with ADHD. This includes focus groups with key stakeholders (Define), extended formative usage evaluation (Refine), and an open preliminary feasibility trial and usability testing (Pilot). Our goal is to develop and preliminary test an online platform that increases engagement, skills generalization, and family involvement in an empirically-supported organization skills intervention for adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Youth ages of 11 to 14 that are attending a participating school
2. referred by school mental health provider as a youth with apparent ADHD-related problems
3. ≥6 symptoms (item score ≥2) of Inattention or Hyperactivity-Impulsivity on the pooled parent and teacher Vanderbilt ADHD Rating Scale
4. ≥3 on the Impairment Rating Scale by parent and teacher (cross-situational impairment)
5. Parent consent and youth assent must be provided

Exclusion Criteria:

1. No presence of conditions that are incompatible with this study's treatment including: Parent or adolescent report of a prior diagnosis of either Autism Spectrum Disorder, Bipolar Disorder, a Dissociative Disorder, Severe visual or hearing impairment, severe language delay or intellectual impairment, or a Psychotic Disorder will be excluded. Rationale: Individuals with these disorders often have very dysregulated behavior and impairments that deviate from the focus of this study.
2. Adolescent is in all-day special education classes or if core classes not in regular education classrooms. Rationale: The vast majority of adolescent with ADHD are served in regular education classrooms and students in full-day self-contained classrooms often have different challenges than students in regular education.
3. Adolescent planning to change (start or stop) psychotropic medication. Note: Adolescents taking medication will be required to meet all entry criteria, including impairment criteria, thus indicating a need for the intervention. Adolescent taking medication for attention or behavior are eligible as long as their medication regimens are stable. Participating parents will also need to be able to read/speak English because all measures are in English, and the intervention will be conducted in English.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
Vanderbilt ADHD Diagnostic Rating Scales (VADRS) Parent Version | Change from Baseline (month 0) to Immediate Post-Intervention (up to 12 weeks later) and 6-months Post-Intervention
  The Vanderbilt scales are DSM-based with teacher- and parent-report forms (Wolraich et al., 1998, 2003). The 18 ADHD symptom items on the Vanderbilt have excellent internal consistency reliability, Cronbach's alpha >.90, and high concurrent validity with other instruments (see Wolraich et al., 2003). Items are rated from 0 (Never) to 3 (Very Often) and the total ADHD severity score range from 0 to 54 with higher scores representing presence of greater parent-rated symptom severity. The present study will examine change in ADHD symptom severity from baseline/pre-intervention (month 0) to post intervention (up to 12 weeks later), and 6-months post-intervention follow-up.
Vanderbilt ADHD Diagnostic Rating Scales (VADRS) Teacher Version | Change from Baseline (month 0) to Immediate Post-Intervention (up to 12 weeks later) and 6-months Post-Intervention
  The Vanderbilt scales are DSM-based with teacher- and parent-report forms (Wolraich et al., 1998, 2003). The 18 ADHD symptom items on the Vanderbilt have excellent internal consistency reliability, Cronbach's alpha >.90, and high concurrent validity with other instruments (see Wolraich et al., 2003). Items are rated from 0 (Never) to 3 (Very Often) and the total ADHD severity score range from 0 to 54 with higher scores representing presence of greater parent-rated symptom severity. The present study will examine change in ADHD symptom severity from baseline/pre-intervention (month 0) to post intervention (up to 12 weeks later), and 6-months post-intervention follow-up.
Impairment Rating Scale (IRS) Parent Version | Change from Baseline (month 0) to Immediate Post-Intervention (up to 12 weeks later) and 6-months Post-Intervention
  The IRS (7-items) was developed to assess the areas of functioning that typically characterize youth with ADHD and is effective in discriminating between youth with and without ADHD (Fabiano et al., 2006). All items are rated from 0 (No Problem) to 6 (Extreme Problem), with higher scores indicating higher levels parent-rated of functional impairment. The present study will examine change in functional impairment levels from baseline/pre-intervention (month 0) to post intervention (up to 12 weeks later), and 6-months post-intervention follow-up.
Impairment Rating Scale (IRS) Teacher Version | Change from Baseline (month 0) to Immediate Post-Intervention (up to 12 weeks later) and 6-months Post-Intervention
  The IRS (7-items) was developed to assess the areas of functioning that typically characterize youth with ADHD and is effective in discriminating between youth with and without ADHD (Fabiano et al., 2006). All items are rated from 0 (No Problem) to 6 (Extreme Problem), with higher scores indicating higher levels teacher-rated of functional impairment. The present study will examine change in functional impairment levels from baseline/pre-intervention (month 0) to post intervention (up to 12 weeks later), and 6-months post-intervention follow-up.
System Usability Scale | Month 6, Month 10, Month 12, Month 18
  10-item technology agnostic scale assessing technology product usability. The total SUS score ranges from 0 to 100, with higher scores indicating higher usability. SUS scores above 80 indicated good usability. The SUS has high internal consistency (α=.91) and high convergent validity with a separate rating of usability and user satisfaction (r=.8). The present study will assess change system usability at the end of software development (month 6), during the intervention trial (month 10), at post-treatment (month 12), and at 6-months post-intervention follow-up (month 18).

SECONDARY OUTCOMES:
Barkley Deficits in Executive Functioning Scale (BDEFS-CA) | Change from Baseline (month 0) to Immediate Post-Intervention (up to 12 weeks later) and 6-months Post-Intervention
  The BDEFS-CA (Barkley, 2012) is measure of children's daily life executive functioning normed on a representative sample of youth. The BDEFS-CA will be collected from parents and adolescents to evaluate the major components of executive functioning.
Behavioral Inhibition System/ Behavioral Activation System, BIS/BAS Scales | Change from Baseline (month 0) to Immediate Post-Intervention (up to 12 weeks later) and 6-months Post-Intervention
  The BIS/BAS Scales (Carver & White, 1994; Pagliaccio et al., 2016) is a 24-item (includes 4 filler items) self-report measure of reinforcement/reward sensitivity rated on a four-point scale to assess theoretical concepts of BIS and BAS function and their roles in motivation, behavior, and affect. Specifically, items on BAS assess pursuit of appetitive goals, reward responsivity, tendencies to seek new, potentially rewarding experiences, and tendencies to act quickly towards goals. Items assessing BIS sensitivity focus more narrowly on concerns about possible negative/punishing events and sensitivity to the occurrence of such events. Higher scores on the BIS and BASC scales indicate greater sensitivity to rewards and punishments. The present study will examine change in reward and reinforcement sensitivity from baseline/pre-intervention (month 0) to post intervention (up to 12 weeks later), and 6-months post-intervention follow-up.
Revised Child Anxiety and Depression Scales (RCADS) | Change from Baseline (month 0) to Immediate Post-Intervention (up to 12 weeks later) and 6-months Post-Intervention
  The RCADS (Chorpita et al., 2005) is a 47-item measure (in the public domain) that assesses adolescent-report of DSM-based anxiety and depression symptoms. The RCADS has been validated for use with students in 3rd through 12th grade. The RCADS has excellent reliability and validity in clinical and school-based samples (Ebesutani et al., 2010). Items are rated from 0 (Never) to 3 (Always), with higher scores indicating higher levels of anxiety and depressive symptoms. The present study will examine change in anxiety and depressive symptom severity from baseline/pre-intervention (month 0) to post intervention (up to 12 weeks later), and 6-months post-intervention follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Research Institute, Washington D.C., District of Columbia, United States